CLINICAL TRIAL: NCT01340495
Title: Pilot Study of Proton Radiation Therapy for Invasive Breast Carcinoma Following Mastectomy
Brief Title: Proton Radiation Therapy for Invasive Breast Cancer Following Mastectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shannon MacDonald, MD, Attending Radiation Oncologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-205
Record Dates: First submitted 2011-04-20; First posted 2011-04-22 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Invasive Breast Cancer
Keywords: Breast Cancer; Mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton Radiation (Experimental): Radiation therapy with proton beam
  Interventions: Radiation: Proton Radiation

INTERVENTIONS:
Radiation: Proton Radiation — 45-50.4 Gy(RBE) to the chest wall and 45-50.5 Gy(RBE) once daily, 5 days per week, for approximately 5 1/2 weeks

SUMMARY:
In this study we are looking at a type of radiation called proton radiation which is known to spare surrounding tissue and organs from radiation. The proton radiation will be delivered using 3D conformal proton radiation or scanned beam/IMPT (Intensity Modulated Proton Radiation Treatment). Proton radiation delivers no dose beyond the region requiring treatment. This may reduce side effects that patients would normally experience with conventional radiation therapy or other means of delivering proton radiation therapy. In this study we are evaluating the effectiveness of using proton radiation delivered to reduce side effects association with radiation treatment.

DETAILED DESCRIPTION:
Proton radiation will be delivered daily for approximately 5 1/2 weeks. Patients will be assessed weekly for any side effects they may be experiencing.

Patients will have follow-up visits 4 weeks after proton therapy ends, at 6 months, 12 months, and then every year for up to five years after treatment. Follow-up visits will include a physical examination, radiological imaging (if necessary), echocardiogram, and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer confined to the breast and regional lymphatics
* Completed mastectomy (complete not partial )breast surgery +/- reconstructive surgery
* Life expectancy > 12 months

Exclusion Criteria:

* Pregnant or breast-feeding
* Prior therapeutic radiation > 200 cGy
* History of a different malignancy unless disease-free for at least 5 years or diagnosed and treated cervical cancer in situ, or basal or squamous cell cancer of the skin
* Prior investigation chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-06; Primary Completion 2017-04 (Actual); Study Completion 2022-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M MacDonald, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Hassan MZO, Awadalla M, Tan TC, Scherrer-Crosbie M, Bakar RB, Drobni ZD, Zarif A, Gilman HK, Supraja S, Nikolaidou S, Zhang L, Zlotoff DA, Hickey SB, Patel SA, Januzzi JL, Keane F, Passeri JJ, Neilan TG, MacDonald SM, Jimenez RB. Serial Measurement of Global Longitudinal Strain Among Women With Breast Cancer Treated With Proton Radiation Therapy: A Prospective Trial for 70 Patients. Int J Radiat Oncol Biol Phys. 2023 Feb 1;115(2):398-406. doi: 10.1016/j.ijrobp.2022.08.036. Epub 2022 Aug 24. PMID 36028065
- [Derived] Jimenez RB, Hickey S, DePauw N, Yeap BY, Batin E, Gadd MA, Specht M, Isakoff SJ, Smith BL, Liao EC, Colwell AS, Ho A, Januzzi JL, Passeri J, Neilan TG, Taghian AG, Lu HM, MacDonald SM. Phase II Study of Proton Beam Radiation Therapy for Patients With Breast Cancer Requiring Regional Nodal Irradiation. J Clin Oncol. 2019 Oct 20;37(30):2778-2785. doi: 10.1200/JCO.18.02366. Epub 2019 Aug 26. PMID 31449469

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proton Radiation
Started | 70
Completed | 69
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Proton Radiation
Number analyzed (Participants) | 70
Age, Continuous [Median (Full Range); unit: years] | 45 [25 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 63
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 63
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 or Higher Radiation Pneumonitis or Any Grade 4 Adverse Event
Description: To determine the feasibility of using proton radiation for the treatment of invasive breast cancer following mastectomy based on the occurrence of grade 3 or > radiation pneumonitis or any grade 4 adverse event within 3 months after the completion of radiation treatment.
Time Frame: From the start of treatment until 3 months after the end of treatment, median duration of treatment of 6 weeks
Population: One participant withdrew from the trial before the start of treatment and was not included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Radiation
Number analyzed (Participants) | 69
Participants | 0

2. Secondary Outcome: The Number of Participants With Acute Skin Toxicities
Description: Summary of the number of participants with any grade acute skin toxicities. Acute skin toxicity was assessed from the start of treatment until 90 days after the end of treatment. Skin toxicity was assessed using Common Terminology Criteria for Adverse Events (CTCAE 4).
Time Frame: From the start of treatment until 3 months after the end of treatment
Population: One participant withdrew from the trial before the start of treatment and was not included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Radiation
Number analyzed (Participants) | 69
Participants | 69

3. Secondary Outcome: Rate and Severity of Radiation Pneumonitis
Description: The number of participants that experienced radiation pneumonitis within three months of the end of treatment. The participants that experienced radiation pneumonitis are grouped by grade. Adverse events were assessed using Common Terminology Criteria for Adverse Events (CTCAE 4).
  * Grade 1: Mild
  * Grade 2: Moderate
  * Grade 3: Severe
  * Grade 4: Life-Threatening
  * Grade 5: Fatal
Time Frame: From the start of treatment until 3 months after the end of treatment and was not included in the analysis population.
Population: One participant withdrew from the trial before the start of treatment and was not included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Radiation
Number analyzed (Participants) | 69
Participants
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0
  Grade 5 | 0

4. Secondary Outcome: Summary of Late Skin Toxicity
Description: A summary of the late skin toxicities experienced by participants. The number of participants effected is shown for each toxicity experienced. Skin toxicities were assessed using Common Terminology Criteria for Adverse Events (CTCAE 4).
Time Frame: From 3 months after the end of treatment up to 5 years
Reporting Status: Not Posted, anticipated posting 2023-01

5. Secondary Outcome: To Evaluate Cosmetic Outcome and Patient Satisfaction With Cosmetic Outcome
Time Frame: From the start of treatment until 5 years post treatment
Reporting Status: Not Posted, anticipated posting 2023-01

6. Secondary Outcome: Acute and Late Toxicity of Breast Reconstruction Following Proton Radiation
Description: Combined summary of the acute (within 3 months of completing treatment) and late (3 months to 5 years after completion of treatment) toxicities experienced by participants thought to be related to breast reconstruction surgery following proton radiation treatment. Toxicities are assessed using Common Terminology Criteria for Adverse Events (CTCAE 4).
Time Frame: From the start of treatment until 5 years post treatment
Reporting Status: Not Posted, anticipated posting 2023-01

7. Secondary Outcome: The Number of Participants That Needed Unplanned Additional Surgery for Breast Reconstruction
Time Frame: From the start of treatment until 5 years post treatment
Reporting Status: Not Posted, anticipated posting 2023-01

8. Secondary Outcome: The Number of Participants With Early Signs of Cardiac Effects From Radiation Therapy
Description: The number of participant that had early signs of cardiac effects from radiation therapy as assessed using a Strain Echo-cardiogram. The data from the Echo-cardiogram was evaluated for signs of negative impacts to cardiac function as determined by the treating physician. Parameters considered in the evaluation of the echo-cardiogram by the physician included myocardial velocity, strain, strain rate, and torsion. Blood-based cardiac bio-markers pro-BNP and ultra-sensitive troponin-I were also assessed. Either a clinically meaningful change in the strain echo-cardiogram parameters or clinically meaningful elevation of the bio-markers was sufficient to be considered to have early signs of cardiac effects.
Time Frame: Baseline and then 4 and 8 weeks post treatment
Population: One participant withdrew from the trial before the start of treatment and was not included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Radiation
Number analyzed (Participants) | 69
Participants | 0

9. Secondary Outcome: Progression Free Survival
Description: Progression-free survival is defined as the duration from the start of radiation to the date of objective disease progression or death due to any cause, whichever is earlier. Disease progression is defined as the appearance of one or more new lesions.
Time Frame: from the start of treatment until the time of disease progression, up to 5 years
Reporting Status: Not Posted, anticipated posting 2023-01

ADVERSE EVENTS:
Time Frame: Weekly during radiation treatment; 1, 2, 6, and 12 months post treatment; then yearly up until 5 years after the end of treatment (median duration of follow-up of about 36 months of follow-up at the time of analysis).
Description: Serious adverse events were defined as adverse events that were serious, life threatening, or fatal and deemed to be at least possibly related to study treatment. Adverse events categorized as 'Other' were grouped together by organ system due to inconsistent terminology used to specify the 'other' adverse event and to highlight overall adverse event trends.
Arm/Group | Proton Radiation
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 20/70
Other Adverse Events (participants affected / at risk) | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Radiation (N=70)
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 (2)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorders - Other, specify (Musculoskeletal and connective tissue disorders) | 7 (10)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 13 (18)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Radiation (N=70)
Abdominal pain (Gastrointestinal disorders) | 16 (28)
Alanine aminotransferase increased (Investigations) | 6 (14)
Alkaline phosphatase increased (Investigations) | 5 (11)
Allergic reaction (Immune system disorders) | 5 (8)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (29)
Anemia (Blood and lymphatic system disorders) | 17 (26)
Anorexia (Metabolism and nutrition disorders) | 7 (8)
Anxiety (Psychiatric disorders) | 28 (97)
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 (110)
Arthritis (Musculoskeletal and connective tissue disorders) | 9 (16)
Aspartate aminotransferase increased (Investigations) | 7 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (67)
Bloating (Gastrointestinal disorders) | 5 (5)
Blurred vision (Eye disorders) | 10 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 13 (21)
Breast pain (Reproductive system and breast disorders) | 17 (37)
Bruising (Injury, poisoning and procedural complications) | 8 (9)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 42 (124)
Chills (General disorders) | 6 (7)
Cognitive disturbance (Nervous system disorders) | 5 (17)
Constipation (Gastrointestinal disorders) | 8 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (35)
Depression (Psychiatric disorders) | 17 (63)
Dermatitis radiation (Injury, poisoning and procedural complications) | 69 (356)
Diarrhea (Gastrointestinal disorders) | 7 (8)
Dizziness (Nervous system disorders) | 13 (22)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (25)
Dysmenorrhea (Reproductive system and breast disorders) | 5 (8)
Dyspareunia (Reproductive system and breast disorders) | 10 (30)
Dysphagia (Gastrointestinal disorders) | 28 (76)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 9 (18)
Fatigue (General disorders) | 67 (459)
Fever (General disorders) | 10 (10)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 39 (101)
Flank pain (Musculoskeletal and connective tissue disorders) | 9 (23)
Flatulence (Gastrointestinal disorders) | 4 (4)
Flu like symptoms (General disorders) | 6 (9)
Fracture (Injury, poisoning and procedural complications) | 6 (9)
Gait disturbance (General disorders) | 7 (12)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 (11)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 5 (10)
Headache (Nervous system disorders) | 18 (40)
Hot flashes (Vascular disorders) | 37 (150)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (16)
Hypertension (Vascular disorders) | 9 (27)
Hypothyroidism (Endocrine disorders) | 4 (13)
Insomnia (Psychiatric disorders) | 19 (46)
Irregular menstruation (Reproductive system and breast disorders) | 6 (12)
Irritability (General disorders) | 4 (10)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 33 (80)
Libido decreased (Psychiatric disorders) | 5 (14)
Lip infection (Infections and infestations) | 4 (5)
Localized edema (General disorders) | 15 (27)
Lung infection (Infections and infestations) | 4 (4)
Lymphedema (Vascular disorders) | 14 (53)
Lymphocyte count decreased (Investigations) | 12 (30)
Menorrhagia (Reproductive system and breast disorders) | 5 (7)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 6 (19)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 48 (214)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (20)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Nausea (Gastrointestinal disorders) | 18 (23)
Neck pain (Musculoskeletal and connective tissue disorders) | 13 (27)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (18)
Pain (General disorders) | 30 (93)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 (77)
Palpitations (Cardiac disorders) | 10 (10)
Paresthesia (Nervous system disorders) | 6 (11)
Pelvic pain (Reproductive system and breast disorders) | 6 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 24 (89)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 39 (106)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 4 (12)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 4 (5)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 6 (8)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 13 (32)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 61 (254)
Skin infection (Infections and infestations) | 14 (21)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 11 (31)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 14 (19)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 7 (11)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 28 (53)
Telangiectasia (Skin and subcutaneous tissue disorders) | 11 (32)
Upper respiratory infection (Infections and infestations) | 12 (17)
Urinary frequency (Renal and urinary disorders) | 5 (5)
Uterine hemorrhage (Reproductive system and breast disorders) | 6 (9)
Vaginal discharge (Reproductive system and breast disorders) | 8 (10)
Vaginal dryness (Reproductive system and breast disorders) | 11 (24)
Vaginal infection (Infections and infestations) | 6 (6)
Vomiting (Gastrointestinal disorders) | 6 (6)
White blood cell decreased (Investigations) | 13 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT01340495/Prot_SAP_ICF_000.pdf